CLINICAL TRIAL: NCT02888379
Title: A Phase 2a, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Safety/Tolerability and Efficacy of TOP1288 200 mg Rectal Solution Once Daily for 4 Weeks in Symptomatic Ulcerative Colitis Patients With Moderate to Severe Disease Activity
Brief Title: Phase 2a Study to Evaluate the Safety/Tolerability and Efficacy of TOP1288 200 mg Rectal Solution Once Daily for 4 Weeks in Ulcerative Colitis
Acronym: TOP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Topivert Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOP1288-TV-02
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TOP1288 200 mg Rectal Solution (Experimental): TOP1288 200 mg Rectal Solution Once Daily for 4 Weeks
  Interventions: Drug: TOP1288
- Placebo Rectal Solution (Placebo Comparator): Placebo (for TOP1288) Rectal Solution Once Daily for 4 Weeks
  Interventions: Drug: Placebo (for TOP1288)

INTERVENTIONS:
Drug: TOP1288
  Arms: TOP1288 200 mg Rectal Solution
Drug: Placebo (for TOP1288)
  Arms: Placebo Rectal Solution

SUMMARY:
A Phase 2a, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Safety/Tolerability and Efficacy of TOP1288 200 mg Rectal Solution Once Daily for 4 Weeks in Symptomatic Ulcerative Colitis Patients with Moderate to Severe Disease Activity

DETAILED DESCRIPTION:
TOP1288, the first in a new class of agents called narrow spectrum protein kinase inhibitors (NSKIs), is being developed as a novel, non-absorbed treatment for ulcerative colitis (UC). UC is a disease of unknown cause characterised by inflammation of the lining of the large intestine and manifesting with abdominal pain and bloody diarrhoea. TOP1288 given rectally has a local anti-inflammatory action in experimental models of UC.

A Phase I placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study of TOP1288 conducted in 61 healthy volunteers demonstrated that rectal administration of TOP1288 at doses up to 200 mg BID for 4 days was safe and well tolerated, with minimal systemic absorption. TOP1288 200 mg, administered once daily, therefore offers the potential for a safe and effective novel approach to treating patients with this serious condition.

This Phase 2a proof-of-concept study will evaluate the 200 mg daily dose of TOP1288, based on its favourable tolerability in the Phase 1 study. It will be administered as TOP1288 200 mg Rectal Solution compared against Placebo Rectal Solution, which contains all non-active excipients present in the active solution. This is a randomised, double-blind, placebo-controlled multicentre study designed to evaluate the safety/tolerability and efficacy of TOP1288 200 mg Rectal Solution following once-daily bedtime treatment for 4 consecutive weeks. The study will include approximately 40 sites in Europe. Randomization to study treatment will be 2:1, with approximately 40 subjects randomised to TOP1288 and approximately 20 subjects randomised to placebo.

The Screening period will be up to 28 days prior to the first day of dosing with double-blind study treatment (Visit 1). A central reading facility will be used to determine eligibility based upon the Screening flexible sigmoidoscopy.

Visit 2 is scheduled for Day 7 of dosing, and Visit 3 for Day 29 of dosing. There will be a 1-week safety follow-up period after Visit 3. The total duration of study participation for a given subject will be up to ~65 days or 9 weeks

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of UC of at least 3 months duration
* Active UC with a Partial Mayo Clinic Score of 4 to 8 at randomization

Key Exclusion Criteria:

* Receiving any rectally administered medication
* Use of biologic agents within 3 months prior to Screening endoscopy
* Use of IV corticosteroids within 4 weeks prior to Screening endoscopy
* Use of oral corticosteroids at a dose >30 mg/day (or budesonide >9 mg/day).
* Patients who have started receiving immune suppressants within 3 months of the Screening endoscopy should not be included.
* Known or suspected pancolitis (unless on oral 5-ASA, steroids or permitted immunomodulators)
* Known or suspected Crohn's disease, indeterminate colitis, microscopic colitis, ischaemic colitis, or radiation-induced colitis, based on medical history, endoscopy, and/or histological findings
* Extensive (>50%) colonic resection or colectomy, or prior history of toxic megacolon within 3 months of Screening
* Patient has active serious infection (e.g., sepsis, pneumonia, abscess) or has had a serious infection (resulting in hospitalisation or requiring parenteral antibiotic treatment) within 6 weeks prior to IMP administration
* Patients testing positive of Clostridium difficile toxin or confirmed with bacterial or parasitical GI infections at Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by the Mayo Clinic modified endoscopic subscore | After 4 consecutive weeks of daily bedtime treatment

SECONDARY OUTCOMES:
Safety as measured by adverse events | To 1 week after the last dose
Safety as measured by vital signs | To 1 week after the last dose
Safety as measured by ECGs | To 1 week after the last dose
Safety as measured by clinical laboratory tests | To 1 week after the last dose
Efficacy as measured by Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score | After 4 consecutive weeks of daily bedtime treatment
Efficacy as measured by Partial Mayo Clinic score (i.e., the sum of the endoscopic, rectal bleeding, and stool frequency subscores) | After 4 consecutive weeks of daily bedtime treatment
Efficacy as measured by endoscopic healing (indicated by the Mayo Clinic modified endoscopic subscore) | After 4 consecutive weeks of daily bedtime treatment
Efficacy as measured by rectal bleeding (indicated by the Mayo Clinic rectal bleeding subscore) | After 4 consecutive weeks of daily bedtime treatment

CONTACTS AND LOCATIONS:
Overall Officials: Simon Travis, FRCP, Principal Investigator — Oxford University Hospitals Trust, John Radcliffe Hospital, Oxford, UK,
Locations (28):
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Czechia (4):
  - Brno
  - Litoměřice
  - Olomouc
  - Prague
- Hungary (7):
  - Budapest
  - Gyöngyös
  - Győr
  - Gyula
  - Szeged
  - Székesfehérvár
  - Vác
- Latvia (2):
  - Daugavpils
  - Riga
- Kaunas, Lithuania
- Poland (6):
  - Bydgoszcz
  - Knurów
  - Skierniewice
  - Sopot
  - Warsaw
  - Wroclaw
- Ukraine (5):
  - Kherson
  - Kyiv
  - Odesa
  - Temopil
  - Zaporizhzhia
- London, United Kingdom